CLINICAL TRIAL: NCT00361309
Title: A Phase II Study of SU011248 in Advanced Hepatocellular Carcinoma
Brief Title: SU011248 in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-348
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: liver cancer; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SU011248 (Experimental): Patients will receive SU011248 37.5 mg/day for 4 weeks continuously followed by 2 weeks of rest per cycle (each cycle = 6 weeks). Patients will be continued on treatment until disease progression, limiting toxicity, or patient withdrawal of consent.
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: SU011248 — Patients will receive SU011248 37.5 mg/day for 4 weeks continuously followed by 2 weeks of rest per cycle (each cycle = 6 weeks).
  Other Names: Sunitinib

SUMMARY:
The main purpose of this study is to begin to collect information and try to learn whether SU011248 works in treating patients with advanced liver cancer. Laboratory studies have shown that SU011248 may block the growth of blood vessels in tumors, which may prevent tumors from growing any further.

DETAILED DESCRIPTION:
* Participants will be given a supply of SU011248 capsules to be taken orally every morning for 4 weeks. After taking SU011248 for 4 weeks, there will be a 2 week rest period when the participant will not take any capsules. This 6-week period is referred to as 1 cycle.
* Participants will continue to receive SU011248 study treatment as long as their disease does not worsen significantly and they are not experiencing any serious side effects.
* During cycle 1 of study treatment, the participant will come to the outpatient clinic once a week for blood work, physical examination and dynamic contrast enhanced magnetic resonance imaging (DCE-MRI), which is done two weeks after they start taking study treatment.
* During cycle two and every cycle thereafter, the participant will be asked to come to the outpatient clinic once every two weeks for physical examination, blood work and urine tests.
* A CT scan or MRI scan to assess the tumor will be performed once during each cycle for the first three cycles, then once every 2 cycles thereafter. ACTH stimulation test will be done every 2 cycles. A MUGA scan may be done at anytime at the discretion of the the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HCC and should have metastatic or locally advanced unresectable disease
* Measurable disease
* 0-1 prior systemic chemotherapy regimens for HCC
* Age 18 years or older
* Life expectancy of greater than 12 weeks
* ECOG performance status of 0-1
* Adequate organ and marrow function
* Women of child-bearing potential must have a negative pregnancy test prior to study entry

Exclusion Criteria:

* Chemotherapy, radiotherapy or major surgery within 4 weeks of study entry
* Receiving any other investigational agents within past 30 days
* Known brain metastases
* CLIP score > 3
* Chronic diarrhea or any disorder that will limit adequate absorption of SU011248
* Prolongation of QTc > 450 msec in screening electrocardiogram or history of familial long QT syndrome
* Uncontrolled intercurrent illness
* Pregnant or lactating women
* Greater than or equal to 2g of protein/24hr

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival of hepatocellular carcinoma (HCC) patients treated with SU011248. | 2 years

SECONDARY OUTCOMES:
Number of adverse events in patients treated with SU011248 for advanced hepatocellular carcinoma | 2 years
Objective Response Rate | 2 years
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew X. Zhu, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Sahani DV, Jiang T, Hayano K, Duda DG, Catalano OA, Ancukiewicz M, Jain RK, Zhu AX. Magnetic resonance imaging biomarkers in hepatocellular carcinoma: association with response and circulating biomarkers after sunitinib therapy. J Hematol Oncol. 2013 Jul 10;6:51. doi: 10.1186/1756-8722-6-51. PMID 23842041